CLINICAL TRIAL: NCT01060670
Title: A Multi-Center, Randomized, Controlled Clinical Trial to Evaluate The Safety and Effectiveness of Integra® Dermal Regeneration Template for the Treatment of Neuropathic Diabetic Foot Ulcers
Brief Title: A Safety and Efficacy Study of INTEGRA® Dermal Regeneration Template for the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRT/DFU US - 2009-3
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Diabetic Ulcer - Foot
Keywords: Foot Ulcer; Diabetic; Wound Healing; Integra Dermal Regeneration Template; Full Thickness; Neuropathic; Omnigraft
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermal Replacement Device (Experimental): Device: INTEGRA® Dermal Regeneration Template
  Interventions: Device: Integra® Dermal Regeneration Template
- Moist Wound Therapy (Active Comparator): 0.9% Saline gel
  Interventions: Other: Conventional Wound Therapy

INTERVENTIONS:
Device: Integra® Dermal Regeneration Template — Application of Integra® Dermal Regeneration Template in diabetic foot ulcer
  Arms: Dermal Replacement Device
Other: Conventional Wound Therapy — Conventional Wound Therapy
  Arms: Moist Wound Therapy

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the INTEGRA® Dermal Regeneration Template for the treatment of diabetic foot ulcers located distal to the malleolus in subjects with diabetes mellitus, neuropathy, and without significantly compromised arterial circulation.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetes mellitus
* Glycosylated hemoglobin, HbA1c, ≤ 12%
* Negative serum pregnancy test at screening for female participants of child-bearing potential
* Willing and able to maintain the required off-loading (as applicable for the location for the ulcer) and applicable dressing changes
* At least one DFU that met the following criteria:

  1. Ulcer was diagnosed as a full-thickness neuropathic DFU that was located distal to the malleolus (excluding ulcers between the toes but including those of the heel),
  2. Minimum 2-cm margin between the qualifying study ulcer and any other ulcers on the specified foot (post debridement),
  3. Area greater than or equal to 1 square centimeter and less than or equal to 12 square centimeters (post debridement at the time of randomization),
  4. Wagner grade 1 or 2,
  5. Depth less than or equal to 5 millimeters with no exposed capsule, tendon or bone and no tunneling, undermining or sinus tracts,
  6. Duration of the study ulcer was at least 30 days at the time of the screening visit
* Adequate vascular perfusion of the affected limb

Exclusion Criteria:

* Suspected or confirmed signs/symptoms of gangrene or wound infection on any part of the limb
* History of hypersensitivity to bovine collagen and/or chondroitin.
* Pregnancy
* Previous treatment under this clinical protocol
* Participation in another clinical trial involving a device or systematically administered investigational study drug or treatment within 30 days of the randomization visit.
* Receiving or scheduled to receive a medication or treatment which, in the opinion of the investigator, was known to interfere with, or affect the rate and quality of wound healing
* Any unstable condition or circumstance that could interfere with treatment regimen compliance
* Excessive lymphedema that could interfere with wound healing
* Unstable Charcot foot or Charcot with boney prominence
* Ulcers secondary to a disease other than diabetes
* Osteomyelitis with necrotic soft bone
* Chopart amputation
* History of bone cancer or metastatic disease of the affected limb, radiation therapy to the foot, or chemotherapy within the 12 months prior to randomization
* Treatment with wound dressings that include growth factors, engineered tissues, or skin substitutes within 30 days of randomization or scheduled to receive such treatment during the study
* Non-study ulcer requiring treatment that could not be treated during the study with moist wound therapy
* History of or intercurrent illnesses or conditions (other than diabetes) that would compromise the safety of the subject, or the normal wound healing process
* Employees or relatives of any member of the investigational site or sponsor
* Size of the study ulcer following debridement decreased by more than 30% during the run in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (32):
  - Costal Clinical Research, Mobile, Alabama
  - Stockdale Podiatry Group, Bakersfield, California
  - Center for Clinical Research, Castro Valley, California
  - Diabetic Foot and Wound Treatment Center, El Centro, California
  - Sacramento Foot and Ankle Center, Fair Oaks, California
  - Advanced Foot Care and Clinical Research Center, Fresno, California
  - Center for Clinical Research, Fresno, California
  - California School of Podiatry Medicine at Samuel Merritt University, Oakland, California
  - Northern California Foot and Ankle Center, Santa Rosa, California
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - South Florida Wound Care Group, Tamarac, Florida
  - C/O Center for Wound Care, Wellington, Florida
  - Village Podiatry Center, Atlanta, Georgia
  - Idaho Falls Infectious Diseases, PLLC, Idaho Falls, Idaho
  - Springfield Clinic, Springfield, Illinois
  - Infectious Disease of Indiana, Indianapolis, Indiana
  - Benchmark Research, Metarie, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Cambridge Health Alliance, Cambridge, Massachusetts
  - Montana Medical Research, Missoula, Montana
  - Advanced Foot and Ankle Center, Las Vegas, Nevada
  - Excelsior Foundation of WNY, Amherst, New York
  - Private Practice, East Setauket, New York
  - Columbia University Medical Center, New York, New York
  - Penn North Center For Advanced Wound Care, Erie, Pennsylvania
  - Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Limb Salvage Center, Dallas, Texas
  - Department of Plastic Surgery, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Foot and Ankle Institute, St. George, Utah
- St. Elisabeth's Hospital, Willemstad, Curacao, Netherlands Antilles

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 36 medical centers between March 2010 and November 2013. The first study participant was enrolled in April 2010 and the last study participant was enrolled in November 2013.
Pre-assignment Details: Participants participated in a Run-In phase that must last a minimum of 14 days, but may have been extended up to 17 days to allow for scheduling of the randomization visit.
Groups:
- Active Treatment: INTEGRA® Dermal Regeneration Template (IDRT) was applied to sharply debrided study ulcer wound bed within an aseptic field. A non-adherent foam dressing, gauze wrap and an offloading/protective device were used in conjunction with the IDRT.
- Control Treatment: Control Treatment was applied to sharply debrided study ulcer wound bed within an aseptic field. Moist wound therapy consisted of 0.9% sodium chloride gel, applied in conjunction with a non-adherent foam dressing, gauze wrap and an offloading/protective device.
Period: Run In
Arm/Group | Active Treatment | Control Treatment
Started | 0 | 545
Completed | 0 | 307
Not Completed | 0 | 238
Not completed — screen failure | 0 | 238
Period: Treatment Phase
Arm/Group | Active Treatment | Control Treatment
Started | 154 | 153
Healed at End of Treatment Phase | 79 | 49
Did Not Heal by Treatment Visit 17 | 49 | 68
Withdrew From Treatment | 26 | 36
Completed | 128 | 117
Not Completed | 26 | 36
Period: Follow up Phase
Arm/Group | Active Treatment | Control Treatment
Started | 128 | 117
Recurrence | 14 | 9
Withdrew From Follow up Phase | 22 | 35
Completed | 106 | 82
Not Completed | 22 | 35

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: INTEGRA® Dermal Regeneration Template (IDRT) was applied to sharply debrided study ulcer wound bed within an aseptic field. A non-adherent foam dressing and a gauze wrap and, an offloading/protective device were to be used in conjunction with the IDRT.
- Control Treatment: Control Treatment consisted of moist wound therapy and was comprised of 0.9% sodium chloride gel, applied in conjunction with a non-adherent foam dressing and a gauze wrap and, an offloading/protective device
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Control Treatment | Total
Number analyzed (Participants) | 154 | 153 | 307
Age, Continuous [Mean (Full Range); unit: years] | 55.8 [31 to 82] | 57.3 [28 to 82] | 56.5 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 118 | 114 | 232
Region of Enrollment [Number; unit: participants]
  United States | 152 | 151 | 303
  Netherlands Antilles | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Complete Wound Closure
Description: 100% closure as assessed by the Investigator and confirmed at 2 consecutive treatment phase visits.
Time Frame: 16 weeks
Population: The results were based on the Investigator assessment and ITT population.
Measure: Number; unit: participants
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 154 | 153
participants | 79 | 49

2. Secondary Outcome: Incidence of Complete Wound Closure
Description: Percentage of subjects with complete wound closure of the study ulcer, as assessed by computerized planimetry, during the treatment phase.
Time Frame: 16 weeks
Population: ITT Population
Measure: Number; unit: percentage of subjects
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 154 | 153
percentage of subjects | 50 | 31

3. Secondary Outcome: Time to Complete Wound Closure
Description: Measures the time to complete wound closure as assessed by the Investigator.
Time Frame: 16 weeks
Population: ITT Population complete wound healed with analyzable data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 79 | 49
days | 52.61 (27.22) | 69.78 (31.73)

4. Secondary Outcome: Time to Complete Wound Closure
Description: Time to complete wound closure, as assessed by computerized planimetry.
Time Frame: 16 weeks
Population: ITT population complete wound healed with analyzable data
Measure: Median (Full Range); unit: days
Groups:
- Dermal Replacement Device: INTEGRA® Dermal Regeneration Template (IDRT) was applied to sharply debrided study ulcer wound bed within an aseptic field. A non-adherent foam dressing, gauze wrap and an offloading/protective device were used in conjunction with the IDRT.
- Moist Wound Therapy: Control Treatment was applied to sharply debrided study ulcer wound bed within an aseptic field. Moist wound therapy consisted of 0.9% sodium chloride gel, applied in conjunction with a non-adherent foam dressing, gauze wrap and an offloading/protective device.
Arm/Group | Dermal Replacement Device | Moist Wound Therapy
Number analyzed (Participants) | 77 | 48
days | 43 [15 to 123] | 78 [8 to 116]

5. Secondary Outcome: Rate of Wound Closure
Description: Rate of wound closure as assessed by computerized planimetry
Time Frame: 16 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage wound closure/week
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 151 | 148
percentage wound closure/week | 7.15 (8.27) | 4.81 (7.34)

6. Secondary Outcome: Incidence of Ulcer Recurrence
Description: Measures the incidence of ulcer recurrence at the site of the study ulcer during the follow up phase.
Time Frame: 12 weeks
Population: ITT Population complete wound healed
Measure: Number; unit: participants
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 79 | 49
participants | 15 | 13

7. Secondary Outcome: Change in Short Form Health Survey (SF-36) Quality of Life Metrics
Description: Short Form Health Survey (SF-36)- Quality of Life Metrics. The SF-36 was utilized and the Physical Function and Bodily Pain subscales were norm-based, with a Mean = 50, SD = 10. Scores could theoretically range from 0 to 100, with higher scores indicating a better health status.
Time Frame: Baseline and 16 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Treatment | Control Treatment
Number analyzed (Participants) | 154 | 153
units on a scale
  Physical Function | 1.28 (11.62) | -1.41 (9.22)
  Bodily Pain | 2.33 (9.42) | -.50 (9.82)

ADVERSE EVENTS:
Time Frame: All events starting after the 1st randomized treatment visit through Follow Up visit 3 will be recorded as AEs.
Arm/Group | Active Treatment | Control Treatment
Serious Adverse Events (participants affected / at risk) | 38/154 | 55/153
Other Adverse Events (participants affected / at risk) | 0/154 | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=154) | Control Treatment (N=153)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
dyspnoea (Cardiac disorders) | 0 (0) | 1 (1)
cataract (Eye disorders) | 0 (0) | 1 (1)
gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
chest pain (General disorders) | 1 (1) | 1 (1)
condition aggravated (General disorders) | 2 (2) | 6 (6)
multi orgain failure (General disorders) | 0 (0) | 1 (1)
non cardiac chest pain (General disorders) | 1 (1) | 0 (0)
cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
abcess (Infections and infestations) | 1 (1) | 0 (0)
abcess limb (Infections and infestations) | 1 (1) | 3 (3)
arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
cellulitis (Infections and infestations) | 7 (7) | 6 (7)
diabetic foot infection (Infections and infestations) | 8 (8) | 6 (7)
gangrene (Infections and infestations) | 0 (0) | 3 (3)
infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
localised infection (Infections and infestations) | 0 (0) | 1 (1)
osteomyelitis (Infections and infestations) | 8 (8) | 15 (15)
perineal abcess (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 3 (3) | 3 (3)
sepsis (Infections and infestations) | 1 (1) | 1 (1)
septic shock (Infections and infestations) | 0 (0) | 1 (1)
soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (3) | 2 (2)
ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
renal hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
convulsion (Nervous system disorders) | 0 (0) | 1 (1)
loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
arterial insufficiency (Vascular disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall not publicly disclose any results/information pertaining to the trial until a multi-center publication is released under sponsor's direction; however, if a multi-center publication is not released within 18 months after completion of analysis of all study data from all studies conducted within the multi center trial, Investigator may publish results at their institution as long as they have given sponsor 30 days to review.